CLINICAL TRIAL: NCT05746624
Title: Procedural Motor Memory in Long COVID-19
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000466; 000466-N
Record Dates: First submitted 2023-02-18; First posted 2023-02-28 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03-27

CONDITIONS: Infectious Metabolic Encephalopathy; Ischemic Stroke; Seizure; Viral Encephalitis, Small and Large Vessel
Keywords: Corona Virus
MeSH Terms: conditions — Ischemic Stroke; Seizures; Encephalitis, Viral; Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Arm 1 Long COVID left handed: Long COVID left handed
  Interventions: Behavioral: keypresses
- Arm 1 Long COVID right handed: Long COVID right handed
  Interventions: Behavioral: keypresses
- Arm 2 Healthy Controls left handed: healthy left handed
  Interventions: Behavioral: keypresses
- Arm 2 Healthy Controls right handed: healthy right handed
  Interventions: Behavioral: keypresses

INTERVENTIONS:
Behavioral: keypresses — benign behavioral intervention-- keypresses

SUMMARY:
Background:

Most people who get COVID-19 seem to recover with no long-term effects. However, some people who recover from acute COVID-19 infections report lingering symptoms. This is called long COVID. Many people with long COVID report symptoms related to the nervous system; these can include problems with fatigue, speech, and memory.

Objective:

To test motor memory in people with long COVID, compared to healthy volunteers.

Eligibility:

People aged 18 to 90 years who are also enrolled in study protocol 000089. Healthy adults are also needed.

Design:

Participants will be screened by telephone. They will confirm they are able to type without discomfort using their nondominant hand. They will confirm they have access to a computer connected to the internet.

All study tasks will be done online. Participants will complete 2 tasks in 2 days.

Participants will be sent a link to a website. The website will give them instructions. They will place the fingers of their nondominant hand over 4 numbers on the keyboard and type a sequence (eg, 4-1-3-2-4). They will type this sequence as often as they can in 10 seconds. Then they will rest for 10 seconds before repeating the task. They will repeat this pattern for 15 minutes.

After they finish the typing task, participants will take a 10-minute questionnaire. They will answer questions about their experiences with COVID-19 and memory issues; they will say which hand they use for tasks such as brushing their teeth or throwing a ball.

Participants will get a notice to repeat the typing task 22 hours after they finish the first one. They should complete the second task within 28 hours....

DETAILED DESCRIPTION:
This study will objectively test procedural motor memory in a group of people with ongoing symptoms following recovery from acute COVID-19 infection.

Primary Objective: We will use a keyboard typing task to investigate procedural memory formation (primary endpoint measure) in the context of COVID-19 infection. We have two

primary comparisons using the same outcome measure

* To compare procedural memory formation between patients with persistent symptoms following COVID-19 infection ( long COVID ) and matched controls who deny symptoms of long COVID (as reported in self-report questionnaires).
* To compare procedural memory formation between long COVID patients with memory complaints and long COVID patients without memory complaints.

Secondary objectives:

Micro-online gains, micro-offline gains, and long-term consolidation (all secondary measures) will be investigated

* between patients with long COVID and matched controls.
* between long COVID patients with memory complaints and long COVID patients without memory complaints

Exploratory objectives: To compare primary and secondary outcome measures between long COVID patients and healthy controls who report prior COVID-19 infection but are not suffering long COVID symptoms

Primary endpoint measure: Early procedural memory formation, as measured by the difference in tapping speed (keypresses/second) between the first and last correct training trial of early learning (first 11 trials) in a keyboard task.

Secondary endpoint measures:

Micro-online learning. Performance improvements within training trials

Micro-offline learning (rapid consolidation). Performance improvements during rest intervals interspersed with training periods.

Longer-term consolidation (24 hours). Performance improvements between the last training trial of Day 1 and the testing trial of Day 2. We hypothesize that early procedural motor memory learning will be reduced in long COVID patients as compared to healthy controls

(primary hypothesis). Seondarily, we hypothesize that micro-online learning, micro-offline learning (rapid consolidation), and longer term consolidation (24 hours) will be also reduced in long COVID patients as compared to controls.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, patient volunteers must meet all of the following criteria:

Ability of subject to understand and the willingness to review an informed consent

Aged at least 18 years at the time of enrollment, and no older than 90 years of age.

Identity of dominant hand

1. Question: Which hand would you choose to hold the pen to write a formal letter?
2. Note: no specific answer is required for inclusion, but it is required for the next question.

English-Speaking:

Ability to type without discomfort using non-dominant hand

Enrolled in the screening phase of Protocol 000089 Post-Coronavirus Disease 19 Convalescence at the National Institutes of Health in the post-COVID convalescence arm (i.e. reports having started recovery from an acute COVID- 19 infection within past six month and is able to provide documentation of a positive COVID-19 PCR or antibody test)

In order to be eligible to participate in this study, healthy volunteers must meet all of the following criteria:

Ability of subject to understand and the willingness to review an acknowledgement of participation agreement

Aged at least 18 years at the time of enrollment, and no older than 90 years of age

English-speaking

Ability to identify dominant hand

1. Question: Which hand would you choose to hold the pen to write a formal letter?
2. Note: no specific answer is required for inclusion, but it is required for the next question.

Ability to type without discomfort using non-dominant hand

Deny active infection with COVID-19, or ongoing symptoms following COVID-19 infection

Ability to use an internet-connected laptop or desktop computer in a private setting located in the continental U.S. to complete the study task.

This protocol can enroll NIH Employees/staff, including NINDS employees/staff. Staff members from our section and their immediate family members are excluded from participation.

EXCLUSION CRITERIA:

Patient group: A patient who meets any of the following criteria will be excluded from participation in this study:

A condition prior to the diagnosis of COVID-19 infection that would significantly confound interpretation of the behavioral task, as determined by the screening clinician (e.g., prior diagnosis of a neurologic condition such as large stroke, Alzheimer s disease or Parkinson s disease, or severe psychiatric condition).

Staff from our section, and their immediate family members

Healthy Volunteer group: A person who meets any of the following criteria will be excluded from participation in this study:

A condition that would significantly confound interpretation of the research tests as determined by the screening clinician (e.g., prior diagnosis of a neurologic condition such as large stroke, Alzheimer s disease or Parkinson s disease, or severe psychiatric condition)

Fever, respiratory symptoms or diagnosis of COVID-19 in the last 14 days.

History of COVID-19 with residual neurologic symptoms following diagnosis that did not resolve within 14 days of disease onset.

Previous participation in this study (platform filter).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with long COVID were recruited from NIH protocol 000089 Post- Coronavirus Disease 19 Convalescence at the National Institutes of Health . These subjects were matched by age and sex to healthy volunteers recruited online using the Prolific.co crowdsourcing platform. All participants were able to review and understand acknowledgment of participation, age 18 at time of enrollment, English-speaking, able to type without discomfort, and with access to a physical keyboard. Healthy volunteers additionally reported not having active fever or residual symptoms following Covid infection.
Sampling Method: Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
To investigate differences in procedural memory formation and consolidation during a keyboard typing task between o patients withpersistent symptoms following COVID- 19 infection ( long COVID )and matched controls who deny symptoms of ... | anticipated to complete data analysis by December 2023
  Early procedural motor memory learning will be measuredby the difference in keypress speed between the first training trial and last correct training trial of the Day 1 typing task.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo G Cohen, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States